Statistical analysis was done in Rstudio version 0.98.501 software with R language. The suitability of variables to normal distribution was examined using analytical methods (Kolmogorov-Smirnov / Shapiro-Wilk tests) in all individuals. Continuous variables were presented with mean ± standard deviation (SD) and classified variables were presented with number-% tables. When all individuals' data values did not show a normal distribution, the Wilcoxon Signed Ranks Test was used for dependent groups. When comparison data levels of D and C groups did not show normal distribution, the Mann-Whitney U test was used for independent groups. Friedman Variance analysis was used for triple comparisons' dependent groups. Food consumption record and food frequency form was analyzed by BEBİS 8.2. Values, where the p-value was below 0.05, were considered statistically significant, and G-Power v. 3.1.7 software was used to determine the number of samples and then generalize to the population.